CLINICAL TRIAL: NCT05038722
Title: Flödescytometrisk utvärdering av Den Blodstillande förmågan Hos Trombocyter Avsedda för Transfusion
Brief Title: Function of Platelets Used for Transfusions
Status: Enrolling by invitation | Type: Observational
Sponsor: Sofia Ramström (Other)
Responsible Party: Sponsor-Investigator, Sofia Ramström, Associated Professor, Örebro University, Sweden
Organization: Örebro University, Sweden (Other)
Other Study IDs: 2020-05968
Record Dates: First submitted 2021-08-24; First posted 2021-09-09 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Thrombocytopenia; Hematologic Malignancy
MeSH Terms: conditions — Thrombocytopenia; Hematologic Neoplasms | interventions — Platelet Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples without DNA retained from the platelet concentrates used for transfusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Platelet transfusion — Transfusion of platelet concentrates according to routine practice.

SUMMARY:
Cytotoxic treatment for malignant hematologic disorders often casue thrombocytopenia that can result in life threatening bleedings. This is prevented by platelet transfusions but these can cause serious transfusion reactions and thus the number of transused platelet concentrates should be limited. It is therefore important that the platelet concentrates contain functional platelets with long circulation time in the bloodstream.

We have developed a method with flow cytometry to measure platelet function markers. It allows us to determine which pathways that are initiated upon activation.

The aim of this project is to assess to what degree spontaneous activation of platelets as well as their activation capacity affects the transfusion response (i.e. uptake in the circulation and circulation time) in the recipient.

The hypothesis is that transfusion of platelets with low spontaneous activation and high activation capacity will lead to a higher transfusion response in the recipient.

DETAILED DESCRIPTION:
Cytotoxic treatment for malignant hematologic disorders often casue thrombocytopenia that can result in life threatening bleedings. This is prevented by platelet transfusions but these can cause serious transfusion reactions and thus the number of transused platelet concentrates should be limited. It is therefore important that the platelet concentrates contain functional platelets with long circulation time in the bloodstream.

The role of platelets in hemostasis is complex. Upon vascular injury, platelets adhere at the injured site where they become activated, release their granule content and aggregate. Activation include changes in receptors, expression of activation markers and become procaoagulant. We have developed a method with flow cytometry to measures these platelet function markers. It allows us to determine which pathways that are initiated upon activation.

Platelets can be stored a maximum of 5-7 days before transfusion. However, the preparation process and subsequent storage can result in platelet lesions, affecting their ability to promote hemostasis and circulate after transfusion.

The aim of this project is to assess to what degree spontaneous activation of platelets as well as their activation capacity affects the transfusion response (i.e. uptake in the circulation and circulation time) in the recipient.

The hypothesis is that transfusion of platelets with low spontaneous activation and high activation capacity will lead to a higher transfusion response in the recipient.

We will be able to examine how this relates to platelet processing methods and storage duration.

Platelets will be transfused on normal indications to participants at the hematology ward. The platelet concentrates choosen to be transfused will be done according to regular routines at the blood center. We will thus not control what concentrates are transfused (i.e. preparation method and storage time) and hence included in the study.

A small sample will be taken from the platelet concentrate shortly before transfusion and platelet function analysed with the flow cytometry method. Transfusion response will be assessed in the participant by calculation of corrected count increment (CCI) which relates the increase in platelet concentration after transfusion to the number of platelets transfused and the blood volume. CCI is calculated at 1 and 24-hours after transfusion. Clincial variables that might affect the transfusion response such as infection and fever will be registered as well as bleeding. The number of days to next platelet transfusion will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* Participant undergoing treatment for malignant hematologic disorders
* Thrombocytopenia
* Require platelet transfusion

Exclusion Criteria:

- Participant requiring HLA-matched platelet transfusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with malignant hematologic disorders undergoing cancer treatment at the Hematology ward.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Corrected count increment (CCI) | 1- and 24 hours after transfusion.
  CCI relates the increase in platelet concentration in participants after transfusion to the number of platelets transfused and the participants blood volume.
Spontaneous and agonist induced expression of platelet activation markers on platelets in platelet concentrates. | Measured on the day of transfusion prior to transfusion.
  Percentage of platelets expressing P-selectin, LAMP-1, phosphatidylserine and the active conformation of fibrinogen receptor.
Spontaneous and agonist induced formation of platelet subpopulations in platelet concentrates. | Measured on the day of transfusion prior to transfusion.
  Percentage of normal sized platelets, small platelets and platelet fragments (microparticles).

SECONDARY OUTCOMES:
Treatment of infection. | Prior to transfusion.
  Use of antibiotics.
Signs of infection - fever. | Prior to transfusion.
  Body temperature measurement.
Bleeding. | Prior to platelet transfusion and 24-hours after the transfusion.
  Signs of bleeding according to WHO-scale (0-4, where 4 is the worst outcome).
Number of platelet transfusions | From beginning of the cytotoxic treatment cycle to inclusion in the study, i.e receiving a study concentrate.
  Total number of platelet transfusions a participant recieved before being incuded in the study (i.e before being transfused with the study specific platelet concentrate) in the treatment cycle.
Days to next platelet transfusion. | After the study platelet concentrate was transfused, followed for up to two weeks after transfusion.
  The number of days until the next platelet transfusion occured after being transfused with the study specific platelet concentrate.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Ramström, Ass. Prof, Principal Investigator — Örebro University, Sweden
Locations (2):
- Sweden (2):
  - Region Östergötland, Linköping
  - Örebro University, Örebro

IPD SHARING:
Plan to Share IPD: Yes
Individual results from flow cytometry analysis of platelet concentrates that underlie results in a publication after deidentification (text, tables and figures).
Time Frame: Starting 6 months after publication, ending 18 months following article publication.
Access Criteria: Researchers who provide a sound methodological proposal in order to achieve aims in the approved proposal. Proposals should be adressed to the principal investigator.